CLINICAL TRIAL: NCT01151670
Title: Use of Pioglitazone for the Prevention of Radiation-Induced Cognitive Dysfunction
Brief Title: Pioglitazone Hydrochloride in Preventing Radiation-Induced Cognitive Dysfunction in Treating Patients With Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00014528; NCI-2009-01452 (Registry Identifier: CTRP); CCCWFU 97409 (Other: Wake Forest University Health Sciences); NCT01586078 (obsolete NCT alias)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Brain Neoplasms, Malignant; Brain Neoplasms, Benign; Malignant Meningioma; Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: radiation therapy; cognitive dysfunction; brain tumor; memory problems; short term memory loss
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Glioblastoma; Astrocytoma; Cognitive Dysfunction; Memory Disorders | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Pioglitazone 22.5 mg once daily by mouth
  Interventions: Drug: pioglitazone
- Arm 2 (Experimental): Pioglitazone 45 mg once daily by mouth
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: pioglitazone — Pioglitazone 22.5 mg daily before, during and after radiation therapy.
  Other Names: Actos
  Arms: Arm I
Drug: Pioglitazone — Pioglitazone 45 mg by mouth daily before, during and after radiation therapy
  Other Names: Actos
  Arms: Arm 2

SUMMARY:
RATIONALE: Pioglitazone hydrochloride may be effective treatment for cognitive dysfunction caused by radiation therapy.

PURPOSE: This phase I trial is studying the side effects and best dose of pioglitazone hydrochloride in preventing radiation-induced cognitive dysfunction in treating patients with brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the tolerability and toxicity associated with two different dose regimens of pioglitazone administered orally as a cytoprotective agent against radiation-induced brain injury.

SECONDARY OBJECTIVE:

I. To evaluate the effect of pioglitazone on glycemic levels and hemoglobin A1c values when pioglitazone is used as a cytoprotective agent concurrent with radiotherapy in normoglycemic patients.

OUTLINE: Patients undergo fractionated external beam radiotherapy, 3-D conformal radiotherapy, or intensity-modulated radiotherapy. Patients receive oral pioglitazone hydrochloride once daily before for 1 week prior to brain irradiation, during and and continuing for 6 months after completion of radiation radiotherapy. After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed brain tumors of the following types: Group 1: malignant brain tumors (glioblastoma multiforme, anaplastic gliomas, brain metastases, and other malignant brain tumors); or Group 2: low grade brain tumors (low grade gliomas, meningiomas, and other low grade brain tumors)
* All stages and grades of brain tumors are eligible
* Patients must have an ECOG performance status of 0-2
* Patients must have agreed to be treated with fractionated, external beam radiation treatment (EBRT) with either curative or palliative intent (the length of the radiation course must at least be ten fractions)
* Patients must have agreed to have CT and MR imaging for purposes of radiation treatment planning, radiation treatment monitoring, and/or radiation treatment evaluation
* Patients must have measurable disease and/or relevant anatomic features using Magnetic Resonance Imaging
* Prior therapies (cytotoxic, surgery, and radiation) are acceptable
* Use of steroids is acceptable when indicated
* Patients must be able to understand and willingly give informed written consent to participate
* Women of childbearing potential must not be pregnant or nursing and must use medically appropriate contraception if sexually active
* Patients must have a life expectancy of greater than 3 months
* Patients must be willing to comply with an oral treatment regimen and be able to swallow oral study tablets

Exclusion Criteria:

* History of allergic reactions to pioglitazone or any other member of the thiazolidinedione family
* Current diagnosis of diabetes as defined by fasting blood sugar > 125, treatment with anti-diabetic medications, or history of diabetes
* Patients who take insulin
* Patients who have NYHA class III or IV heart failure
* Patients who have elevated transaminases (AST or ALT > 2.5 times normal limit)
* Patients who have significantly impaired renal function (creatinine >= 1.5)
* Patients who are significantly anemic (hematocrit < 33% in men, or < 30% in women)
* Patients who have symptomatic edema (>= grade 2)
* Patients who are on medications that have been shown to have a drug interaction with pioglitazone: atorvastatin (doses > 80 mg/day), systemic anti-fungals, medications with significant CYP 3A4 inhibiting properties
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac, arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study if their pregnancy precludes radiation treatment because ionizing radiation used in radiation treatment is an agent with known potential for teratogenic or abortifacient effects
* Patients with psychiatric or social illnesses that may impair compliance with the trial requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Best tolerated dose of 2 different doses of orally administered pioglitazone | From first dose to 1 day after last dose of drug

SECONDARY OUTCOMES:
Toxicities associated with both dose levels | From first dose to 1 day after last dose of drug
To evaluate the effect of pioglitazone on glycemic levels and hemoglobin A1c values when pioglitazone is used as a cytoprotective agent concurrent with radiotherapy in normoglycemic patients. | From first dose to 1 day after last dose of drug

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chan, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States